CLINICAL TRIAL: NCT02352961
Title: An Implementation Science Study Investigating Profiles of Men Interested in Medical Male Circumcision (MMC), Barriers and Methods to Increase the Uptake of MMC Among Older Men in South Africa
Brief Title: An Implementation Science Study Investigating Profiles of Men Interested in MMC
Acronym: Imbizo
Status: Completed | Type: Observational
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: AUR2-4-121
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Medical Male Circumcision
Keywords: Unrecognised condition

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Exclusive Intervention Strategy — The "Exclusive Intervention Strategy" aimed at men aged 25 - 49 years and "Active Follow-up strategy"

SUMMARY:
There are both supply and demand gaps in our understanding of how best to implement MMC services. In terms of supply of MMC services, there is a need to better understand what the best way is of efficiently accessing mature men(25-49 years old) . The investigators also want to understand the type of service delivery approach and environment that would make mature men(25-49 years old) feel more comfortable when attending an MMC clinic. Demand of MMC requires identifying messaging that works to address mature men's (25-49 years old) issues so that they might be willing to undergo MMC. To further advance HIV prevention and advocacy of male circumcision the investigators also need to consider the perspectives of women on what approach MMC messaging should take. A combination of male and female viewpoints could inform MMC outreach messaging where IEC materials are tailored to address the barriers to MMC. Identifying the specific barriers to MMC among males and including the perspectives

DETAILED DESCRIPTION:
Part I (Formative Period) Given these issues, in addition to establishing a baseline estimate of the ages and risk behaviours of males currently undergoing MMC at the Aurum clinic over a six month period, we include a qualitative research component. We conducted research in 2014 to establish a baseline estimate of the ages and risk behaviours of males undergoing MMC at the Aurum clinic over a six month period. The baseline estimate (Ethics reference number M130711) will be referred to as the formative Part I. The formative Part I includes a quantitative and qualitative research component. The qualitative component will include both genders and be used to develop MMC recruitment messaging tailored to mature men(25-49 years old) . Men will provide their opinion on circumcision and on what type of marketing message they feel will encourage mature men (25-49 years old) to be circumcised. Women will also provide their perspectives on male circumcision and what messaging could be used to encourage their partners or male family members to be circumcised. During this study, we explored if women have a role in promoting male circumcision to their partners, family and the community. These qualitative findings will be used to develop interventions to increase the ratio of men (25-49 years old) mature, or at least of higher risk men, undergoing MMC at the clinic. These interventions and the outcomes related to them will be presented as an amendment to this protocol after the baseline and qualitative data are collected and analysed.

Part II (Intervention Period) Findings from the formative period will be used to develop interventions to increase the ratio of men (25-49 years)mature, or at least of higher risk men, undergoing MMC at the clinic. During this proposed intervention period we would like to evaluate the effectiveness of those interventions and the outcomes related to them. These proposed interventions will directly address the barriers to MMC that challenge uptake of MMC among mature men (25-49 years). Additionally, epidemiologic research will be conducted among men attending our MMC clinic to evaluate whether mature men (25-49 years) exhibit, as is presumed, higher risk profiles for HIV. We will also explore the cost-effectiveness of this strategy.

ELIGIBILITY:
Inclusion Criteria for Cross Sectional Component Inclusion Criteria:

All males who meet the following criteria will be eligible for inclusion:

* Are aged 18 years or older (no upper age limit)
* Have never been completely medically circumcised (as opposed to partial circumcision)
* Willing and able to give their written informed consent so that the information collected during the clinic visit can be analysed for research purposes.

Inclusion Criteria Qualitative Component for males

All males who meet the following criteria will be eligible for inclusion:

* Present at Aurum's male circumcision clinic during the cross sectional component or men who indicate no interest in medical male circumcision
* Are between the ages of 25 and 49 inclusive
* Are not circumcised at the time of the interview as assessed through visual examination
* Is willing and able to provide written informed consent.
* Willing for the qualitative session to be tape recorded

Inclusion Criteria for Qualitative Component for females Women who meet the following criteria will be eligible for inclusion

* Are 18 and above (no upper age limit)
* Has a partner who is participating in the cross sectional component, is not in a relationship but lives in the vicinity of Ekurhuleni North district or is part of a women's organization within the community where the clinic is located
* Is willing and able to provide written informed consent
* Willing for the qualitative session to be tape recorded

Inclusion Criteria Part II (Intervention Period) Inclusion Criteria for the "Exclusive Intervention Strategy" Men who meet the following criteria will be eligible for inclusion in the intervention period

* Are between the ages 25 and 49 years inclusive
* Has never been medically circumcised
* Is willing and able to provide written informed consent

Inclusion Criteria for the "Active Follow-up Intervention" Men who meet the following criteria will be eligible for inclusion

* Are between the ages 25 and 49 years inclusive
* Has never been medically circumcised
* Is willing and able to provide written informed consent
* Has contra-indication/s to MMC on the day of presentation for MMC
* Is willing to provide contact information for retention

Exclusion Criteria for all Aims:

* Men who are unable to communicate sufficiently (in English or local languages) to complete medical forms and/or research questionnaires for the cross sectional component.
* Men and women who do not in the opinion of staff obtaining consent have the capacity to provide written informed consent will be excluded from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males 18 and above accessing medical male circumcision services in Ekurhuleni North, South Africa
  Females 18 and above who live in the vicinity of Ekurhuleni North, South Africa
Sampling Method: Non-Probability Sample
Enrollment: 2817 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Current proportion of mature men (25-49 years) presenting for and undergoing MMC | 6 months
  To describe the current proportion of mature men (25-49 years) presenting for and undergoing MMC compared to all men (18 and above) during a 6 month period when routine service delivery and outreach messaging will be employed at one Aurum site.
Particular barriers to MMC among men (25-49 years) | 6 months
  To describe the particular barriers to MMC among men (25-49 years) regardless of circumcision status, develop tailored messaging and outreach materials promoting MMC to mature men.
Barriers to MMC and using the perspective of women | 6 months
  To investigate the particular barriers to MMC and using the perspective of women develop tailored messaging and outreach materials promoting MMC to mature men.
Effectiveness of offering an "Exclusive Intervention Strategy" | 6 months
  Evaluate the effectiveness of offering an "Exclusive Intervention Strategy" comprised of customized services to mature (25-49 years) men. To achieve this aim we will compare the proportion of mature men (25-49 years) presenting for MMC during the formative and intervention periods.

SECONDARY OUTCOMES:
Risk behaviours | 6 months
  Identify risk behaviours (e.g. multiple partners; inconsistent condom use and STI symptoms) of men currently presenting at the Aurum MMC clinic.
Compare risk behaviours to national prevalence | 6 months
  Compare risk behaviours of men presenting for MMC with that of national prevalence estimates of risk behaviour.
Risk profile, age and source of recruitment | 6 months
  Describe the risk profile, age and sources of recruitment of men presenting at the clinic. To achieve this aim we will examine each of these factors over time.
Factors associated with the intervention | 6 months
  Identify whether the intervention is associated with HIV risk behaviours (for example multiple partners), having adjusted for age. This is to identify if the intervention has resulted in men attending for MMC with a different risk profile over and above any anticipated age differences.
Socio-demographic factors | 6 months
  Identify socio-demographic factors associated with HIV risk behaviours, among mature men (25-49 years).
Effectiveness of active follow-up | 6 months
  Evaluate the effectiveness of an active follow-up system on completion of MMC among mature men (25-49 years) who present for MMC but who are initially referred for care due to contra-indication to MMC
Cost effectiveness | 6 months
  To determine the cost-effectiveness of this intervention among mature men (25-49 years).

CONTACTS AND LOCATIONS:
Overall Officials: Salome Charalambous, MBBCH, PhD, Principal Investigator — Aurum Institute
Locations (1):
- The Aurum Institute, Gauteng, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Publications will be shared and made available

REFERENCES:
- [Derived] Chetty-Makkan CM, Grund JM, Muchiri E, Price MA, Latka MH, Charalambous S. High risk sexual behaviours associated with traditional beliefs about gender roles among men interested in medical male circumcision in South Africa. AIDS Res Ther. 2021 Jun 22;18(1):33. doi: 10.1186/s12981-021-00359-7. PMID 34158082
- [Derived] Grund JM, Chetty-Makkan CM, Ginindza S, Munyai R, Kisbey-Green H, Maraisane M, Charalambous S. Effectiveness of an "Exclusive Intervention Strategy" to increase medical male circumcision uptake among men aged 25-49 years in South Africa. BMC Public Health. 2018 Jul 13;18(1):868. doi: 10.1186/s12889-018-5729-6. PMID 30005663